CLINICAL TRIAL: NCT01658592
Title: Deep Brain Stimulation of the Nucleus Accumbens and the Ventral Anterior Internal Capsule as a Novel Treatment in Severe Alcohol Addiction
Brief Title: Deep Brain Stimulation of the Nucleus Accumbens and the Ventral Anterior Internal Capsule for Severe Alcohol Addiction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guodong Gao (Other)
Collaborators: Tang-Du Hospital (Other)
Responsible Party: Sponsor-Investigator, Guodong Gao, Neurosurgery Department, Tang-Du Hospital
Organization: Tang-Du Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: NAc-VC DBS for alcohol addict
Record Dates: First submitted 2012-07-26; First posted 2012-08-07 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-08

CONDITIONS: Addiction
Keywords: Alcohol Addiction;; Deep Brain Stimulation;; Nucleus Accumbens;; Ventral Anterior Internal capsule;
MeSH Terms: conditions — Behavior, Addictive; Alcoholism | interventions — Deep Brain Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- NAC-VC Deep Brain Stimulation (Experimental): The contractors located in NAc and VC are ON at the same time
  Interventions: Other: Deep brain stimulation; Other: Placebo
- Placebo A (Sham Comparator): Stimulator setting is OFF
  Interventions: Other: Deep brain stimulation; Other: Placebo
- Placebo B (Experimental): The contractor located in NAc is on
  Interventions: Other: Deep brain stimulation; Other: Placebo
- Placebo C (Experimental): The contactor located in VC is on
  Interventions: Other: Deep brain stimulation; Other: Placebo

INTERVENTIONS:
Other: Deep brain stimulation — Stimulator setting is ON
Other: Placebo — Stimulator setting is OFF

SUMMARY:
The main objective of this study is to assess the efficacy of bilateral deep brain stimulation (DBS) of the nucleus accumbens (NAc) and the ventral anterior internal capsule (VC) as a novel treatment in severe alcohol addiction. The included patients have been treated so far with drugs that inhibits alcohol, or psychological behavior training.

Our hypothesis is that bilateral NAc-VC DBS will significantly reduce the craving for alcohol and thus enable the patients to decrease their alcohol intake substantially.

DETAILED DESCRIPTION:
The nucleus accumbens (NAc) is considered associating with addiction. The ventral anterior internal capsule(VC) is proved a effective target to obsessive compulsive disorder(OCD). Like other addiction behaviors most alcohol addicts contain obsessive compulsive symptom. We explored an operation method, that is, in the Leksell stereotactic positioning system take VC as the point of entry, take NAc as the point of target, then make sure that the distance between entry and target points are included in the four contacts of electrode of DBS. When stimulator is ON the investigators can adjust parameters so that the coverage of electrode contains both Vc and NAc. The investigators suppose that bilateral NAc-VC DBS will significantly reduce the craving for alcohol and thus enable the patients to decrease their alcohol intake substantially.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Long lasting alcohol addiction (fulfilled diagnostic-criteria according to DSM-IV,ICD-10)
* At least one detoxication-treatment without a long-term period of abstinence has already taken place
* Long-term inpatient treatment to support abstinence have occurred
* Free patient's decision / Informed Consent (existing comprehensive ability in meaning, methodology and execution of the study and ability of acceptance)
* If prior medication, stable dosage of psychopharmacological drugs over the last three months, which shall, after checking be retained during the study

Exclusion Criteria:

* Hospitalization for psychotic symptoms
* Clinical relevant psychiatric comorbidity (such as schizophrenic psychoses, bipolar affective diseases, severe personality disorder, and so on. And diagnosed by criteria according to DSM-IV,ICD-10)
* Contraindications of a MRI-examination, e.g. implanted cardiac pacemaker/ heart defibrillator
* Current and in the last six months existent paranoid-hallucinated symptomatology
* Foreign aggressiveness in the last six months
* Verbal IQ < 85 (evaluated with the Wechsler Adult Intelligence Scale- Chinese Revised (WAIS-CR)
* Stereotactic respectively neurosurgical intervention in the past
* Other neurological diseases
* Contraindications of a stereotactic operation, e.g. increased bleeding-disposition, cerebrovascular diseases (e.g. arteriovenous malfunction, aneurysms, systemic vascular diseases)
* Serious and instable organic diseases (e.g. instable coronal heart disease)
* tested positively for HIV
* pregnancy and/or lactation

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2012-07; Primary Completion 2014-03 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Reduction of Alcohol | 7 months
  Reduction of the dosage of alcohol(all kinds of liquor were converted into pure alcohol) comparing baseline and the particular ward rounds during and at the end of the crossover-design.

SECONDARY OUTCOMES:
Craving | 7 months
  10-point visual analog scale (VAS) of craving

OTHER OUTCOMES:
Psychological components | 7 months
  Addiction severity(ASI); Psychological components (Anxiety (BAI-21 item); Depression (BDI-21 item); Quality of life (WHOQL-Brief); Health condition(SF-36).

CONTACTS AND LOCATIONS:
Overall Officials: Gao G Dong, Doctor, Principal Investigator — Department of neurosurgery, Tangdu Hospital
Locations (1):
- Department of neurosurgery, Tangdu Hospital, Xi'an, Shaanxi, China